CLINICAL TRIAL: NCT04380753
Title: A Phase 1, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of AMG 510 in Subjects of Chinese Descent With Advanced/Metastatic Solid Tumors With KRAS p.G12C Mutation (CodeBreaK 105)
Brief Title: AMG 510 Ethnic Sensitivity Study (CodeBreaK 105).
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20190147
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Advanced/Metastatic Solid Tumors With KRAS p.G12C Mutation
Keywords: AMG510 phase 1; Chinese Descent; Advanced Solid Tumors; KRAS p.G12C Mutation
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects will be enrolled and will receive AMG 510 PO QD.
  Interventions: Drug: AMG 510

INTERVENTIONS:
Drug: AMG 510 — Subjects will be enrolled and will receive AMG 510 PO QD.

SUMMARY:
To evaluate safety, tolerability, PK, and preliminary efficacy of AMG 510 PO QD in subjects of Chinese descent with KRAS p.G12C-mutant advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects greater than or equal to 18 years old
* Subject is of Chinese ancestry
* Pathologically documented, advanced/metastatic solid tumor with KRAS p.G12C mutation identified

Exclusion Criteria:

* Active brain metastases from non-brain tumors.
* Myocardial infarction within 6 months of study day 1.
* Gastrointestinal (GI) tract disease causing the inability to take oral medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2026-06-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- Hong Kong (2):
  - University of Hong Kong, Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin, New Territories
- Taiwan (2):
  - Veterans General Hospital - Taichung, Taichung
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants were enrolled in the study in Hong Kong and Taiwan. The study is currently ongoing; results are reported up to the primary data cut-off date of 31 December 2021.
Pre-assignment Details: Administration of sotorasib orally (PO) once daily (QD) was permitted to continue until there was evidence of disease progression, intolerance to study medication, or withdrawal of consent. The primary analysis occurred after all participants enrolled had the opportunity to complete 6 months on study or withdrew from study.
Groups:
- Sotorasib: Participants received Sotorasib 960 mg PO QD until there was evidence of disease progression, intolerance to study medication, or withdrawal of consent.
Period: Overall Study
Arm/Group | Sotorasib
Started | 12
Completed | 6
Not Completed | 6
Not completed — Participants continuing study | 4
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all enrolled participants who received at least 1 dose of sotorasib.
Arm/Group | Sotorasib
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: DLTs were defined as any of the following adverse events (AEs) where a relationship to sotorasib could not be ruled out.
  Hematological toxicity
  * febrile neutropenia
  * neutropenic infection
  * grade 4 neutropenia
  * grade ≥ 3 thrombocytopenia for > 7 days
  * grade 3 thrombocytopenia with grade ≥ 2 bleeding
  * grade 4 thrombocytopenia
  * grade 4 anemia.
  Non-hematological toxicity
  * grade ≥ 4 vomiting or diarrhea
  * grade 3 diarrhea or grade 3 vomiting lasting more than 3 days despite optimal medical support
  * grade ≥ 3 nausea for 3 days or more despite optimal medical support
  * any other grade ≥ 3 adverse event.
Time Frame: Day 1 to Day 21
Population: DLT analysis set: DLT-evaluable subjects (participants who either experienced a DLT or did not experience a DLT but received at least 80% of the planned doses of investigational product within the 21-day DLT window) in the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotorasib
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: Number of Participants With Treatment-emergent AEs (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. A TEAE was defined as an AE starting on or after first dose of study treatment.
  Treatment-related TEAEs were any TEAEs considered related to investigational product by the investigator. If relationship was missing, the event was assumed treatment-related.
  Clinically significant changes from the participant's baseline values in vital signs, 12-lead electrocardiograms, and clinical laboratory safety tests were reported as AEs.
Time Frame: Day 1 until the end of study (or primary data cut-off date for ongoing participants); median [min, max] duration was 5.57 [1.5, 13.7] months
Population: Safety analysis set: all enrolled participants who received at least 1 dose of sotorasib.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotorasib
Number analyzed (Participants) | 12
Participants
  Any TEAEs | 11
  Any Treatment-related TEAEs | 4

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sotorasib
Description: Pharmacokinetic (PK) parameters were determined from the concentration-time profile using standard non-compartmental approaches and considering the profile over the complete sampling interval.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Days 1 and 8
Population: PK analysis set: all participants who received at least 1 dose of sotorasib and had at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sotorasib
Number analyzed (Participants) | 12
ng/mL
  Day 1 | 9010 (5200)
  Day 8 | 6330 (3030)

4. Primary Outcome: Time to Achieve Cmax (Tmax) of Sotorasib
Description: PK parameters were determined from the concentration-time profile using standard non-compartmental approaches and considering the profile over the complete sampling interval.
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Days 1 and 8
Population: PK analysis set: all participants who received at least 1 dose of sotorasib and had at least 1 PK sample collected.
Measure: Median (Full Range); unit: hours
Arm/Group | Sotorasib
Number analyzed (Participants) | 12
hours
  Day 1 | 0.85 [0.50 to 6.00]
  Day 8 | 0.96 [0.47 to 5.90]

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24h) of Sotorasib
Description: as for outcome 4
Time Frame: Pre-dose and 0.25, 0.5, 1, 2, 4, 6, and 24 hours post-dose on Days 1 and 8
Population: PK analysis set: all participants who received at least 1 dose of sotorasib and had at least 1 PK sample collected.
Measure: Mean (Standard Deviation); unit: hours*ng/mL
Arm/Group | Sotorasib
Number analyzed (Participants) | 12
hours*ng/mL
  Day 1 | 73200 (43700)
  Day 8: number analyzed (Participants) | 11
  Day 8 | 37400 (32000)

6. Secondary Outcome: Objective Response (OR)
Description: Measured by computed tomography (CT) or magnetic resonance imaging (MRI). Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines.
Time Frame: Day 1 until the end of study (approximately 12 months)
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Duration of Response (DoR)
Description: Measured by CT or MRI. Assessed per RECIST version 1.1 guidelines.
Time Frame: Day 1 until the end of study (approximately 12 months)
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Progression-free Survival (PFS)
Description: Measured by CT or MRI. Assessed per RECIST version 1.1 guidelines.
Time Frame: Day 1 until the end of study (approximately 12 months)
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Disease Control Rate (DCR)
Description: Measured by CT or MRI. Assessed per RECIST version 1.1 guidelines.
Time Frame: Day 1 until the end of study (approximately 12 months)
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Time to Response (TTR)
Description: Measured by CT or MRI. Assessed per RECIST version 1.1 guidelines.
Time Frame: Day 1 until the end of study (approximately 12 months)
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Duration of Stable Disease
Description: Measured by CT or MRI. Assessed per RECIST version 1.1 guidelines.
Time Frame: Day 1 until the end of study (approximately 12 months)
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Day 1 until the end of study (or primary data cut-off date for ongoing participants); median [min, max] duration was 5.57 [1.5, 13.7] months
Description: Safety analysis set: all enrolled participants who received at least 1 dose of sotorasib.
Arm/Group | Sotorasib
All-Cause Mortality (participants affected / at risk) | 2/12
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sotorasib (N=12)
Ileus (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Liver function test abnormal (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sotorasib (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Euthyroid sick syndrome (Endocrine disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Mucosal inflammation (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Xerosis (General disorders) | 1
Herpes simplex (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Weight increased (Investigations) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin mass (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-09-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT04380753/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT04380753/SAP_001.pdf